CLINICAL TRIAL: NCT00638313
Title: A Phase 1, Placebo-Controlled, Randomized Study To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Following Single, Escalating Subcutaneous Doses Of PF-04603629 In Type 2 Diabetic Adult Subjects
Brief Title: Single-Dose Study Of PF-04603629 In Type 2 Diabetic Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: B0571001
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2009-07-31 (Estimated); Status verified 2008-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — PF 04603629

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- PF-04603629 (Experimental)
  Interventions: Biological: PF-04603629

INTERVENTIONS:
Biological: Placebo — Subjects will be given either Placebo or PF-04603629.
  Arms: Placebo
Biological: PF-04603629 — Subjects will be given either Placebo or PF-04603629. The specific dose of PF-04603629 given depended on the Cohort to which the patient was assigned. Doses administered ranged from 1 mg to 70 mg.
  Arms: PF-04603629

SUMMARY:
PF 04603629 is a long acting exendin proposed for the treatment of Type 2 diabetes mellitus. The purpose of this study is to characterize the safety, tolerability, pharmacokinetics and glucose lowering capabilities following a single subcutaneous dose.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Hb A1c lower or equal to 11%

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Evidence of diabetic complications with significant end-organ damage

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-08; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To characterize the pharmacokinetics of PF-04603629 in serum after administration, under fasted conditions, of single, escalating, subcutaneous doses of PF-04603629 to adult subjects with T2DM. | 1 week per dose group
To characterize the pharmacodynamic effect (glucose AUC lowering) of single, escalating, subcutaneous doses of PF-04603629 administered to adult subjects with T2DM. | 1 week per dose group
To evaluate the safety and tolerability of escalating, single subcutaneous doses of PF-04603629 administered to adult subjects with T2DM. | 1 week per dose group

SECONDARY OUTCOMES:
No secondary outcomes listed in the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0571001&StudyName=Single-Dose%20Study%20Of%20PF-04603629%20In%20Type%202%20Diabetic%20Subjects